CLINICAL TRIAL: NCT05561972
Title: Assessment of the Efficacy Of Multifractional Intercalated Hyaluronic Acid Injection for Genitourinary Syndrome of Menopause Using 3D High Frequency Vaginal Ultrasound
Brief Title: The Ultrasonographic Assessment of Efficacy of Injectable Hyaluronic Acid for Genitourinary Syndrome of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/900/87
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Genitourinary Syndrome of Menopause; Sexual Function Disturbances
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: injectable multifractional intercalated hyaluronic acid [Armonia®, Regenyal, Italy] — Armonia® 2 ml was injected into the vaginal wall with a standardized injection technique called Cannulated Intravaginal Injection Technique®. In this technique, Armonia® was injected as drops at 40 different points on the entire vaginal wall using 8 different entry points

SUMMARY:
Genitourinary syndrome of menopause (GSM) is a definition including vaginal dryness, burning, vaginal pruritus, dyspareunia and urinary symptoms which can have a negative effect on women's sexuality and quality of life. The most common strategies to overcome GSM are non-hormonal (vaginal lubricants, topical moisturizers, energy-based devices etc.) and hormonal therapies. While vaginal lubricants are used during sexual intercourse and have temporary effects on vaginal epithelium, vaginal moisturizers are "bio-adhesive" products that can improve vaginal atrophy symptoms when used regularly. These products have not serious side effects but long-term effectiveness is not established. In the last decade, energy-based devices like laser and radiofrequency were used for treatment of GSM. Nevertheless, side effects and safety problems associated with these methods lead to uncertainty about the use of these methods in GSM therapy. Local and systemic estrogen therapies have been widely used for decades, but there is limited data on the persistence of the effect after estrogen use is stopped.

Hyaluronic acid (HA) is a glycosaminoglycan molecule that is an essential element of the extracellular matrix, with water-retention properties and regulatory effects on inflammation, scarring, and angiogenesis]. To date, many studies reported short-term improving effects of topical HA on GSM symptoms and have used subjective assessment of sexual symptoms and vaginal health scoring tools to investigate the effect of vaginal use of topical HA. However, since the injection of HA into the vagina will have a direct effect on the vaginal epithelium, it would be reasonable to expect a longer efficacy on GSM symptoms.

The methods used to diagnose GSM are subjective or provide unreliable objective evidence. Recently demonstrated as an objective diagnostic tool for GSM, 3D high frequency vaginal ultrasound (3D-HFVU) was used to separately measure anterior vaginal wall (ant-VWT) and posterior vaginal wall thickness (post-VWT) in contrast to 2D ultrasonography. To date, there are no studies to evaluate the effect of HA injection on the vaginal epithelium ultrasonographically.

The aim of the study was to investigate the effect of multifractional intercalated HA (MIC-HA) [Armonia®, Regenyal, Italy] injection on ant-VWT and post-VWT using 3D-HFVU, and also to assess the relationship between sexual functions and VWT increase in women with GSM after the injection. This is the first study to assess the effect of vaginal injection of MIC-HA on ant-VWT and post-VWT separately using 3D-HFVU.

ELIGIBILITY:
Inclusion Criteria:Postmenopausal women who had vaginal irritation, burning, vaginal pruritus, dryness and dyspareunia -

Exclusion Criteria:The presence of pelvic organ prolapse greater than stage I, vulvovaginitis, genital carcinoma, previous vaginal surgery, current use of vaginal moisturizers or lubricants, local or systemic estrogen treatment and antidepressant use, women those with known hypersensitivity to hyaluronic acid, betadine or lidocaine

-

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline anterior and posterior vaginal wall thickness at 4 weeks as detected by 3D high-frequency endovaginal ultrasound | The baseline and 4 weeks after intervention

SECONDARY OUTCOMES:
Turkish version of the Female Sexual Function Index | The baseline and 4 weeks after intervention

OTHER OUTCOMES:
Vaginal health index | The baseline and 4 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No